CLINICAL TRIAL: NCT00423319
Title: A Phase 3 Randomized, Double-blind, Active-controlled, Parallel-group, Multi-center Study to Evaluate the Safety and Efficacy of Apixaban in Subjects Undergoing Elective Total Hip Replacement Surgery (The Advance-3 Study Apixaban Dosed Orally Versus Anticoagulation With Injectable Enoxaparin to Prevent Venous Thromboembolism)
Brief Title: Study of an Investigational Drug for the Prevention of Thrombosis-related Events Following Hip Replacement Surgery (ADVANCE-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-035
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Prevention of deep vein thrombosis and; pulmonary embolism after total hip replacement surgery
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban, 2.5 mg BID plus placebo (Active Comparator): Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
  Interventions: Drug: Apixaban; Drug: Enoxaparin-matching placebo
- Enoxaparin, 40 mg QD plus placebo (Experimental): Participants received enoxaparin, 40 mg QD subcutaneously, and matching apixaban-placebo tablets BID
  Interventions: Drug: Enoxaparin; Drug: Apixaban-matching placebo

INTERVENTIONS:
Drug: Enoxaparin — Subcutaneous, 40 mg, once daily, 5 weeks
  Other Names: Lovenox®
  Arms: Enoxaparin, 40 mg QD plus placebo
Drug: Apixaban — Oral tablets, 2.5 mg, twice daily, 5weeks
  Other Names: BMS-562247; Eliquis®
  Arms: Apixaban, 2.5 mg BID plus placebo
Drug: Enoxaparin-matching placebo — Administered as injection
  Arms: Apixaban, 2.5 mg BID plus placebo
Drug: Apixaban-matching placebo — Administered as oral tablets
  Arms: Enoxaparin, 40 mg QD plus placebo

SUMMARY:
The purpose of this study is to learn whether apixaban can prevent the blood clots in the leg (deep vein thrombosis) and lung (pulmonary embolism) that sometimes occur after hip replacement surgery and to learn how apixaban compares with enoxaparin in preventing these clots. The safety of apixaban will also be studied

ELIGIBILITY:
Key Inclusion Criteria

* Patients undergoing elective unilateral total hip replacement or a revision of at least 1 component of a total hip replacement.
* Patients who were willing and able to undergo bilateral ascending contrast venography
* Either sex, any race, 18 years and older

Key Exclusion Criteria

* Known or suspected bleeding or coagulation disorder in the patient or his or her first-degree relative
* Known or suspected history of heparin-induced thrombocytopenia
* Known coagulopathy
* Active bleeding or at high risk for bleeding
* Brain, spinal, ophthalmologic, or major surgery or trauma within the past 90 days
* Active hepatobiliary disease
* Alcohol and/or substance abuse within the past year
* Any condition for which surgery or administration of an anticoagulant is contraindicated
* Two consecutive blood pressure readings within 15 to 30 minutes with supine systolic blood pressure >180 mm Hg or supine diastolic blood pressure >105 mm Hg
* Clinically significant laboratory abnormalities at the enrollment visit:
* Hemoglobin <10 g/dL
* Platelet count <100,000/mm^3
* Creatinine clearance <30 mL/min, as estimated by the method of Cockcroft and Gault
* Alanine aminotransferase or aspartate aminotransferase >2*upper limit of normal or a total bilirubin ≥ 1.5*1 (unless an alternative causative factor such as Gilbert's syndrome was identified)
* Need for ongoing treatment with a parenteral or oral anticoagulant (eg, subjects with mechanical valves, warfarin eligible atrial fibrillation)
* Current use of dextrans or fibrinolytics
* Treatment with medications affecting coagulation or platelet function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5407 (Actual)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (122):
- United States (19):
  - Capstone Clinical Trials, Inc, Birmingham, Alabama
  - West Alabama Research, Llc, Birmingham, Alabama
  - Martin Bowen Hefley Orthopedics, Little Rock, Arkansas
  - Orthoarkansas, P.A., Little Rock, Arkansas
  - Uc Davis Medical Center, Sacramento, California
  - Colorado Orthopedic Consultants, Pc, Aurora, Colorado
  - Advanced Orthopedic And Sports Medicine Specilists, Denver, Colorado
  - Denver-Vail Orthopedics, P.C., Denver, Colorado
  - Pab Clinical Research, Brandon, Florida
  - Research Alliance, Inc., Clearwater, Florida
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Phoenix Clinical Research, Llc, Tamarac, Florida
  - Atlanta Knee And Sports Medicine, Decatur, Georgia
  - Americana Orthopedics, Boise, Idaho
  - Bosie Orthopedic Clinic, Meridian, Idaho
  - University Orthopedic Center, Altoona, Pennsylvania
  - Gill Orthopedic Center, Lubbock, Texas
  - Robert R. King, Md, Lubbock, Texas
  - Unlimited Research, San Antonio, Texas
- Argentina (4):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Monte Grande, Buenos Aires
- Australia (9):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Southport, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Windsor, Victoria
  - Local Institution, Perth, Western Australia
- Belgium (5):
  - Local Institution, Antwerp
  - Local Institution, Brasschaat
  - Local Institution, Genk
  - Local Institution, Hasselt
  - Local Institution, Leuven
- Canada (15):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ajax, Ontario
  - Local Institution, Cambridge, Ontario
  - Local Institution, Chatham, Ontario
  - Local Institution, Guelph, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, St. Catharines, Ontario
  - Local Institution, Stratford, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- China (4):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Qingdao, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
- Denmark (7):
  - Local Institution, Amager
  - Local Institution, Frederiksberg
  - Local Institution, Herlev
  - Local Institution, Hvidovre
  - Local Institution, Hørsholm
  - Local Institution, København NV
  - Local Institution, Silkeborg
- France (4):
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Saint-Etienne
  - Local Institution, Saint-Saulve
- Germany (3):
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt am Main
  - Local Institution, Rheinfelden
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Kecskemét
  - Local Institution, Szeged
  - Local Institution, Szolnok
- India (5):
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Ludhiana, Punjab
  - Local Institution, Lucknow, Uttar Prsdesh
  - Local Institution, Bangalore
  - Local Institution, Mangalore
- Israel (5):
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Kfar Saba
  - Local Institution, Ẕerifin
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Ciudad Madero, Tamaulipas
- Norway (5):
  - Local Institution, Gjettum
  - Local Institution, Kongsvinger
  - Local Institution, Lillehammer
  - Local Institution, Tynset
  - Local Institution, Tønsberg
- Poland (5):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Romania (2):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
- Russia (6):
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Yaroslavl
- Spain (2):
  - Local Institution, Badalona-Barcelone
  - Local Institution, Barcelona
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm
- Ukraine (6):
  - Local Institution, Cherkassy
  - Local Institution, Chernivtsy
  - Local Institution, Dnipropetrovsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kyiv
  - Local Institution, Sevastopol
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Wigan, Lancashire
  - Local Institution, Epsom, Surrey

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Pineo GF, Gallus AS, Raskob GE, Chen D, Ramirez LM, Ramacciotti E, Lassen MR, Wang L. Apixaban after hip or knee arthroplasty versus enoxaparin: efficacy and safety in key clinical subgroups. J Thromb Haemost. 2013 Mar;11(3):444-51. doi: 10.1111/jth.12109. PMID 23279103
- [Derived] Lassen MR, Gallus A, Raskob GE, Pineo G, Chen D, Ramirez LM; ADVANCE-3 Investigators. Apixaban versus enoxaparin for thromboprophylaxis after hip replacement. N Engl J Med. 2010 Dec 23;363(26):2487-98. doi: 10.1056/NEJMoa1006885. PMID 21175312

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5765 subjects were enrolled, and 5407 were randomized to double-blind study drug.
Period: Overall Study
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Started | 2708 (Randomized) | 2699 (Randomized)
Participants Who Received Treatment | 2673 | 2659
Completed | 2484 | 2447
Not Completed | 224 | 252
Not completed — Death | 2 | 0
Not completed — Adverse Event | 93 | 112
Not completed — Withdrawal by Subject | 86 | 99
Not completed — Lost to Follow-up | 4 | 3
Not completed — Poor compliance or noncompliance | 1 | 1
Not completed — No longer meets study criteria | 15 | 15
Not completed — Other | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo | Total
Number analyzed (Participants) | 2708 | 2699 | 5407
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.79) | 60.6 (11.82) | 60.8 (11.81)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 1608 | 1605 | 3213
  65 to younger than 75 years | 770 | 767 | 1537
  75 years and older | 330 | 327 | 657
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1430 | 1451 | 2881
  Male | 1278 | 1248 | 2526
Region of Enrollment [Number; unit: Participants]
  United States | 450 | 441 | 891
  Spain | 32 | 29 | 61
  Ukraine | 217 | 219 | 436
  Russian Federation | 274 | 276 | 550
  Israel | 57 | 56 | 113
  United Kingdom | 77 | 78 | 155
  India | 56 | 56 | 112
  France | 75 | 74 | 149
  Hungary | 152 | 150 | 302
  Mexico | 73 | 74 | 147
  Canada | 359 | 356 | 715
  Argentina | 53 | 54 | 107
  Belgium | 59 | 60 | 119
  Poland | 184 | 185 | 369
  Romania | 24 | 25 | 49
  Australia | 101 | 99 | 200
  Denmark | 99 | 99 | 198
  Germany | 135 | 134 | 269
  Norway | 47 | 48 | 95
  China | 121 | 124 | 245
  Sweden | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Rate of Composite of Adjudicated Venous Thromboembolic Event (VTE)-Related (Pulmonary Embolism and Symptomatic and Asymptomatic Deep Vein Thrombosis[DVT]) and All-cause Death During the Intended Treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. A mandatory bilateral ascending contrast venogram was to be obtained on Day 35 (± 3). Patients with confirmed symptomatic DVT at any time, or asymptomatic DVT upon venography, were to receive treatment for DVT according to the investigator's standard of care. Signs and symptoms suggestive of VTE included, but were not limited to: 1) lower extremity DVT: erythema, warmth, pain, swelling, tenderness; and 2) PE: pleuritic chest pain, dyspnea, cough, hemoptysis, syncope, light-headedness/dizziness, tachypnea, and tachycardia. Intended Treatment Period started on day of randomization and, for patients who received treatment, ended at the later of 2 days after last dose of study drug or 38 days after the first dose (presurgery) of study drug. For randomized patients who did not receive study drug, the period ended 38 days after randomization.
Time Frame: Day 1 (first dose of study drug) to later of 2 days after last dose or 38 days after first dose
Population: All randomized participants who, during the Intended Treatment Period, had an adjudicated and evaluable bilateral venogram, had an adjudicated venous thromboembolic event, or died of any cause.
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 1949 | 1917
Percentage of events/patients evaluated | 1.39 [0.95 to 2.02] | 3.86 [3.08 to 4.83]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p < 0.0001, Farrington-Manning test — Statistically significant at the 1-sided 0.025 level; Risk Ratio (RR) = 0.36, 95% CI 2-sided [0.22 to 0.54] — Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p < 0.0001, Farrington-Manning test — Statistically significant at the 1-sided 0.025 level; Risk Difference = -2.47, 95% CI 2-sided [-3.54 to 1.50] — Apixaban-enoxaparin

2. Secondary Outcome: Rate of Composite of Adjudicated Proximal Deep Vein Thrombosis (DVT), Nonfatal Pulmonary Embolism, and Venous Thromboembolic Event-related Death With Onset During Intended Treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. Each patient was categorized as having no proximal DVT, having proximal DVT, being nonevaluable for proximal DVT, having no distal DVT, having distal DVT, or being nonevaluable for distal DVT. Adjudication criteria were: Normal=All deep veins were visualized, and there was no intraluminal filling defect (ILFD). ILFD=An area of reduced, or absent filling, at least partially surrounded with contrast medium in ≥ 2 projections or a lack of filling in a vessel in which there was a cut-off that had the configuration of a thrombus. Indeterminate=A lack of filling of a region of the deep vein system, proximal or distal, without the presence of an ILFD elsewhere in the same region. Not Done=A venography was not performed. Proximal DVT was found if any of the proximal veins had an ILFD. Pulmonary embolism was radiographically (angiography, V/Q scan, computed tomography) determined.
Time Frame: Day 1 (first dose of study drug) to later of 2 days after last dose or 38 days after first dose
Population: Randomized participants with either an adjudicated event or an adjudicated evaluable bilateral venogram
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2199 | 2195
Percentage of events/patients evaluated | 0.45 [0.24 to 0.85] | 1.14 [0.77 to 1.69]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p < 0.0001, Farrington-Manning test — Statistically significant at the 1-sided 0.025 level; Risk Ratio (RR) = 0.40, 95% CI 2-sided [0.15 to 0.80] — Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p = 0.0054, Chi-squared — Statistically significant at the 1-sided 0.025 level; Risk difference = -0.68, 95% CI 2-sided [-1.27 to -0.17] — Apixaban-enoxaparin

3. Secondary Outcome: Rates of Adjudicated All-cause Death, VTE-related Death, Pulmonary Embolism (PE), Nonfatal PE, Deep Vein Thrombosis (DVT) (Symptomatic and Asymptomatic), Symptomatic and Asymptomatic Proximal and Distal DVT During the Intended Treatment Period
Description: VTE=venous thromboembolic event; VTE-related death=combination of fatal or nonfatal PE and symptomatic or asymptomatic DVT. Event rate=Number of events divided by the number of patients evaluated.
Time Frame: Day 1 (first dose of study drug) to later of 2 days after last dose or 38 days after first dose
Population: All participants randomized to treatment
Measure: Number; unit: Percentage of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2708 | 2699
Percentage of events/patients evaluated
  All-cause death | 0.11 | 0.04
  VTE-related death | 0.04 | 0.00
  PE (fatal or nonfatal) | 0.11 | 0.19
  Nonfatal PE | 0.07 | 0.19
  All DVT (n=1944, 1911) | 1.13 | 3.56
  Symptomatic DVT | 0.04 | 0.19
  Asymptomatic DVT (n=1943, 1907) | 1.08 | 3.30
  Proximal DVT (n=2196, 2190) | 0.32 | 0.91
  Distal DVT (1951, 1908) | 1.03 | 2.99
  Symptomatic proximal DVT | 0.04 | 0.15
  Asymptomatic proximal DVT (n=2195, 2187) | 0.27 | 0.73
  Symptomatic distal DVT | 0.04 | 0.04
  Asymptomatic distal DVT (n=1950, 1907) | 0.97 | 2.94

4. Secondary Outcome: Rate of Major Bleeding, Clinically Relevant Nonmajor Bleeding (CRNM), Major or CRNM, and Any Bleeding During the Treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. Major bleeding event defined as a bleeding event that was 1) Acute clinically overt bleeding accompanied by at least 1 of the following: decrease in hemoglobin of ≥ 2 g/dL over a 24-hour period, transfusion of ≥2 units of packed red blood cells; bleeding that occurred in at least 1 of the following sites: intracranial, intra-spinal, intraocular, pericardial, an operated joint and requires reoperation or intervention, intramuscular with compartment syndrome, or retroperitoneal; 2) Fatal. CRNM was defined as acute clinically overt bleeding that did not satisfy the criteria for a major bleeding event and met at least 1 of the following: epistaxis, gastrointestinal bleed, hematuria, bruising/ecchymosis, or hemoptysis. Minor bleeding was defined as an acute clinically overt bleeding event that did not meet the criteria for major bleeding or a CRNM. Fatal bleeding event was defined as bleeding that was the primary
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluted
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Percentage of events/patients evaluted
  Major bleeding | 0.82 [0.54 to 1.25] | 0.68 [0.42 to 1.08]
  CRNM | 4.08 [3.39 to 4.90] | 4.51 [3.79 to 5.38]
  Major or CRNM | 4.83 [4.08 to 5.71] | 5.04 [4.27 to 5.94]
  Any bleeding | 11.71 [10.55 to 12.99] | 12.56 [11.36 to 13.88]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p = 0.54, Chi-squared — 2-sided P-Value; Difference in event rates = 0.15, 95% CI 2-sided [-0.33 to 0.64] — Major bleeding. Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p = 0.43, Chi-squared — 2-sided P-Value; Difference in event rates = -0.44, 95% CI 2-sided [-1.53 to 0.66] — CRNM. Apixaban-enoxaparin
Statistical Analysis 3: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p = 0.72, Chi-squared — 2-sided P-Value; Difference in event rates = -0.21, 95% CI 2-sided [-1.38 to 0.95] — Major or CRNM. Apixaban-enoxaparin
Statistical Analysis 4: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; p = 0.34, Chi-squared — 2-sided P-Value; Difference in event rate = -0.85, 95% CI 2-sided [-2.61 to 0.90] — Any bleeding. Apixaban-enoxaparin

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Bleeding Adverse Events (AEs), and Death as Outcome
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. All suspected bleeding events were to be reported by the investigator as either an AE or SAE and adjudicated by the Independent Central Adjudication Committee (ICAC). Definitions of bleeding outcomes: Acute clinically overt bleeding =new onset, visible bleeding, or signs or symptoms suggestive of bleeding with confirmatory imaging techniques that could detect the presence of blood.
Time Frame: First dose of study drug (presurgery) through 30 days after the last dose of study drug
Population: All participants who received at least 1 dose of study medication
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  SAEs | 18 | 18
  Bleeding AEs | 15 | 21
  Death | 2 | 0

6. Secondary Outcome: Number of Participants With a Bleeding-related Adverse Event During the Treatment Period
Description: All suspected bleeding events were to be reported by the investigator as either an adverse event or serious adverse event or and adjudicated by the Independent Central Adjudication Committee (ICAC). Definitions of bleeding outcomes: Acute clinically overt bleeding =new onset, visible bleeding, or signs or symptoms suggestive of bleeding with confirmatory imaging techniques that could detect the presence of blood. All acute clinically overt bleeding events were adjudicated by the ICAC as a major bleeding event or a clinically relevant nonmajor bleeding event; suspected minor bleeding events were not sent for adjudication.
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Postprocedural hematoma | 20 | 23
  Operative hemorrhage | 19 | 14
  Incision site hematoma | 14 | 10
  Incision site hemorrhage | 13 | 19
  Postprocedural hemorrhagic | 4 | 7
  Hematuria traumatic | 1 | 1
  Periorbital hematoma | 1 | 0
  Subcutaneous hematoma | 1 | 0
  Traumatic hematoma | 0 | 1
  Hematoma | 34 | 38
  Wound hemorrhage | 18 | 15
  Hemorrhage | 13 | 13
  Hematuria | 41 | 39
  Hemorrhage urinary tract | 1 | 1
  Urethral hemorrhage | 0 | 2
  Epistaxis | 33 | 25
  Hemoptysis | 3 | 1

7. Secondary Outcome: Number of Participants With a Bleeding-related Adverse Events During the Treatment Period (Continued)
Description: as for outcome 6
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Bloody discharge | 16 | 13
  Catheter site hemorrhage | 6 | 5
  Injection site hemorrhage | 4 | 10
  Injection site hematoma | 3 | 28
  Infusion site hematoma | 1 | 0
  Vessel puncture site hematoma | 1 | 0
  Hematocrit decreased | 18 | 21
  Red blood cell count decreased | 14 | 20
  Blood urine present | 8 | 6
  Blood urine | 1 | 1
  Occult blood positive | 1 | 0
  Fibrin D dimer increased | 0 | 1
  Hematochezia | 6 | 2
  Mallory-Weiss Syndrome | 4 | 0
  Hematemesis | 3 | 2
  Melaena | 3 | 1
  Rectal hemorrhage | 3 | 1
  Gingival bleeding | 2 | 3
  Anal hemorrhage | 1 | 0
  Diarrhea hemorrhagic | 1 | 0
  Diverticulum intestinal hemorrhagic | 1 | 0
  Gastrointestinal hemorrhage | 1 | 1
  Intra-abdominal hematoma | 1 | 0
  Duodenal ulcer hemorrhage | 0 | 1
  Hemorrhoidal hemorrhage | 0 | 1
  Mouth hemorrhage | 0 | 1

8. Secondary Outcome: Number of Participants With a Bleeding-related Adverse Event During the Treatment Period (Continued)
Description: as for outcome 6
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Groups:
- Apixiban, 2.5 mg BID Plus Placebo: Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
Arm/Group | Apixiban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Hemorrhagic anemia | 20 | 15
  Ecchymosis | 5 | 9
  Petechiae | 2 | 2
  Hemorrhage subcutaneous | 1 | 0
  Increased tendency to bruise | 0 | 5
  Vaginal hemorrhage | 2 | 0
  Menorrhagia | 1 | 0
  Uterine hemorrhage | 0 | 1
  Conjunctival hemorrhage | 1 | 0
  Hematoma infection | 1 | 0
  Spinal hematoma | 0 | 1

9. Secondary Outcome: Number of Participants With Neurologic Adverse Events With Onset During the Treatment Period
Description: Neurologic events were based on Medical Dictionary for Regulatory Activities search categories.For new or worsening events that were not related to the site of surgery, additional information was collected on a specific form. In addition, neurology consultation was to be obtained for these patients.
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Paraesthesia | 32 | 19
  Hypoaesthesia | 29 | 35
  Burning sensation | 7 | 5
  Peroneal nerve palsy | 5 | 6
  Hypotonia | 4 | 4
  Dysarthria | 3 | 1
  Paresis | 2 | 1
  Cervicobrachial syndrome | 1 | 1
  Coordination abnormal | 1 | 0
  Hypertonia | 1 | 1
  Neuropathy peripheral | 1 | 2
  Peripheral nerve lesion | 1 | 1
  Radiculitis | 1 | 0
  Paralysis | 0 | 1
  Muscular weakness | 7 | 11
  Nerve injury | 2 | 1
  Femoral nerve injury | 1 | 0
  Sciatic nerve injury | 1 | 0
  Peroneal nerve injury | 0 | 1
  Diplopia | 1 | 0
  Gait disturbance | 1 | 0

10. Secondary Outcome: Number of Participants With Marked Abnormalities (MA) in Clinical Laboratory Test Results During the Treatment Period
Description: preRx=predose; LLN=lower limit of normal; ULN=upper limit of normal. MA criteria: Hemoglobin: >2 g/dL decrease from preRx or value ≤ 8 g/dL; hematocrit (%): <0.75*preRx; platelet count (*10^9 cells/L): <100,000/mm^3; erythrocytes (*10^6 cells/μL): <0.75*preRx level; leukocytes (*10^3 cells/μL): < 0.75*LLN or >1.25*ULN, or if preRx LLN use < 0.8*preRx or >ULN if preRx >ULN use >1.2*preRx or <LLN; basophils (*10^3 cells/μL): >400/mm^3; eosinophils (*10^3 cells/μL): > 0.75*10^3 cells/μL; lymphocytes (*10^3 cells/μL): >0.75*10^3 cells/μL; monocytes (*10^3 cells/μL): >2000/mm^3; neutrophils (*10^3 cells/μL): <1.0;
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Hemoglobin, low (n=2605, 2587) | 2189 | 2218
  Hematocrit, low (n=2554, 2536) | 1274 | 1350
  Platelet count, low (n=2597, 2576) | 6 | 9
  Erythrocytes, low (n=2558, 2540) | 1310 | 1377
  Leukocytes, low (n=2632, 2617) | 54 | 54
  Leukocytes, high (n=2632, 2617) | 385 | 360
  Basophils (absolute), high (n=2629, 2613) | 1 | 3
  Eosinophils (absolute), high (n=2629, 2613) | 75 | 70
  Lymphocytes (absolute), low (n=2629, 2613) | 383 | 382
  Lymphocytes (absolute), high (n=2629, 2613) | 3 | 3
  Monocytes (absolute), high (n=2629, 2613) | 9 | 11
  Neutrophils (absolute), low (n=2629, 2613) | 5 | 4

11. Secondary Outcome: Number of Participants With Marked Abnormalities (MA) in Clinical Laboratory Test Results During the Treatment Period (Continued)
Description: preRx=predose; LLN=lower limit of normal; ULN=upper limit of normal. Alanine aminotransferase (ALT) (U/L): >3 *ULN: alkaline phosphatase (ALP) (U/L): >2* ULN; aspartate aminotransferase (ASP) (U/L): >3 *ULN; bilirubin, direct (mg/dL): >2*ULN; bilirubin, total (mg/dL): >2*ULN; BUN (mg/dL): >2*ULN; creatinine (mg/dL): >1.5*ULN; calcium (mg/dL): < 0.8*LLN or >1.2 *ULN, or if preRx <LLN use <0.75* preRx or >ULN if preRx >ULN use > 1.25*preRx or <LLN; chloride (mEq/L): <0.9*LLN or >1.1*ULN, or if preRx <LLN use <0.9*preRx or >ULN if preRx >ULN use >1.1* preRx or <LLN; bicarbonate (mEq/L): < 0.75* LLN or >1.25*ULN, or if preRx <LLN use <0.75*preRx or >ULN if preRx >ULN use >1.25*preRx or <LLN; potassium (mEq/L): < 0.9*LLN or >1.1*ULN, or if preRx <LLN use <0.9*preRx or >ULN if preRx >ULN use >1.1* preRx or < LLN; sodium (mEq/L): <0.95* LLN or >1.05×ULN, or if preRx <LLN use <0.95* predose or >ULN if preRx >ULN use >1.05 *preRx or < LLN.
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Alkaline phosphatase, high (n=2631, 2618) | 55 | 57
  Alanine aminotransferase, high (n=2629, 2616) | 50 | 83
  Aspartate aminotransferase, high (n=2629, 2616) | 73 | 73
  Bilirubin, direct, high (n=2622, 2604) | 145 | 139
  Bilirubin, total, high (n=2630, 2617) | 24 | 12
  Blood urea nitrogen (BUN), high (n=2618, 2598) | 19 | 17
  Creatinine, high (n=2618, 2598) | 21 | 25
  Calcium, total, low (n=2618, 2598) | 7 | 18
  Calcium, total, high (n=2618, 2598) | 0 | 1
  Chloride, serum, low (n=2615, 2594) | 6 | 6
  Bicarbonate, low (n=2615, 2595) | 8 | 8
  Potassium, serum, low (n=2614, 2594) | 73 | 73
  Potassium, serum, high (n=2614, 2594) | 61 | 47
  Sodium, serum, low (n=2615, 2594) | 29 | 23
  Sodium, serum, high (n=2615, 2594) | 5 | 4

12. Secondary Outcome: Number of Participants With Marked Abnormalities (MA) in Clinical Laboratory Test Results During the Treatment Period (Continued)
Description: preRx=predose; LLN=lower limit of normal; ULN=upper limit of normal. Glucose, fasting (mg/dL): <.8*LLN or >1.5*ULN, or if preRx <LLN use <.8*preRx or >ULN if preRx >ULN use >2*preRx or <LLN; protein, total (g/L): If missing preRx use ≥2, or if value ≥4 or preRx =0 or .5 use ≥2, or if preRx=1 use ≥3, or if preRx =2 or 3 use ≥4; creatine kinase (U/L): >5*ULN; uric acid (mg/dL): >.5* ULN, or if preRx >ULN use >2*preRx; blood, urine: If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx =2 or 3 use ≥4; glucose, urine : If missing preRx use ≥2, or if value ≥4, or if preRx=0 or .5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4; RBC, urine (hpf): If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx dose= 1 use ≥3, or if preRx=2 or 3 use ≥4; WBC, urine (h): If missing preRx use ≥2, or if value ≥4, or if preRx =0 or .5 use ≥2, or if preRx =1 use ≥3, or if preRx=2 or 3 use ≥4.
Time Frame: First dose of study drug (presurgery) through 2 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Glucose, fasting serum, high (n=14, 17) | 0 | 1
  Protein, total, low (n=2618, 2596) | 747 | 752
  Protein, total, high (n=2618, 2596) | 3 | 1
  Creatine kinase, high (n=2630, 2616) | 615 | 642
  Uric acid, high (n=2618, 2597) | 2 | 3
  Blood, urine, high (n=2588, 2568) | 275 | 234
  Glucose, urine, high (n=2588, 2568) | 68 | 76
  Leukocyte esterase, urine, high (n=21, 41) | 0 | 4
  Protein, urine (n=2588, 2568) | 169 | 168
  Red blood cells (RBC), urine, high (n=1310, 1230) | 216 | 173
  White blood cells (WBC),urine, high (n=1311, 1228) | 217 | 229

13. Secondary Outcome: Number of Participants With Adverse Events Related to Elevations in Liver Function Test Results With Onset During the Treatment Period
Description: Treatment guidelines were provided for jaundice and elevated results of liver function tests.
Time Frame: First dose of study drug (presurgery) through 30 days after the last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Participants
  Aspartate aminotransferase increased | 48 | 67
  Alanine aminotransferase increased | 40 | 61
  Gamma-glutamyltransferase increased | 27 | 54
  Blood bilirubin increased | 17 | 7
  Bilirubin conjugated increased | 11 | 12
  Hepatic enzyme increased | 9 | 16
  Liver function test results abnormal | 4 | 9
  Transaminases increased | 1 | 1
  Cholelithiasis | 2 | 0
  Hepatitis toxic | 2 | 0
  Cholecystitis acute | 1 | 0
  Cholestasis | 1 | 0
  Hyperbilirubinemia | 1 | 0
  Postcholecystectomy syndrome | 1 | 0
  Cholecystitis | 0 | 1
  Hepatic pain | 0 | 1
  Hepatitis | 0 | 1
  Hepatomegaly | 0 | 1
  Jaundice cholestatic | 0 | 1
  Hypoalbuminemia | 0 | 1
  Hypoproteinemia | 0 | 1
  Yellow skin | 0 | 1

14. Secondary Outcome: Rates of Adjudicated Myocardial Infarction (MI)/Stroke, MI, Stroke, and Thrombocytopenia During the Intended Treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. All suspected events were reported by investigator. Acute MI=the presence of a clinical situation (eg, abnormal history, physical examination, new electrocardiogram changes) suggestive of an MI and at least 1 of the following: elevated creatine kinase (CK)-MB or troponin T or troponin I ≥2*upper limit of normal (ULN); if CK-MB or troponin values not available, total CK ≥2*ULN; or new significant (≥0.04 sec) Q waves in ≥2 contiguous leads. Stroke=a new focal neurologic deficit of sudden onset lasting at least 24 hours that was not due to a readily identifiable nonvascular cause. Adjudication classified each reported stroke as primary hemorrhagic, nonhemorrhagic, infarction with hemorrhagic conversion, or unknown type. Thrombocytopenia=after 3 days as drop in platelet count to <100,000/mm^3 for patients with a baseline value >150,000/mm^3 or a >50% decline, if the baseline value was ≤150,000/mm^3.
Time Frame: Day 1 (first dose of study drug) to later of 2 days after last dose or 38 days after first dose
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percent of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Number analyzed (Participants) | 2673 | 2659
Percent of events/patients evaluated
  MI/stroke | 0.22 [0.09 to 0.51] | 0.26 [0.12 to 0.56]
  MI | 0.19 [0.07 to 0.46] | 0.11 [0.02 to 0.35]
  Stroke | 0.04 [0.00 to 0.24] | 0.15 [0.05 to 0.41]
  Thrombocytopenia | 0.07 [0.00 to 0.30] | 0.11 [0.02 to 0.35]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; Difference in event rates = -0.04, 95% CI 2-sided [-0.34 to 0.26] — Apixaban-enoxaparin. MI/stroke
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; Difference in event rates = 0.07, 95% CI 2-sided [-0.17 to 0.34] — Apixaban-enoxaparin. MI
Statistical Analysis 3: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; Difference in event rates = -0.11, 95% CI 2-sided [-0.35 to 0.07] — Apixaban-enoxaparin. Stroke
Statistical Analysis 4: Comparison: Apixaban, 2.5 mg BID Plus Placebo vs Enoxaparin, 40 mg QD Plus Placebo; Test type: Superiority or Other; Difference in event rates = -0.04, 95% CI 2-sided [-0.26 to 0.17] — Apixaban-enoxaparin. Thrombocytopenia

ADVERSE EVENTS:
Groups:
- Apixaban, 2.5 mg BID + Placebo: Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
- Enoxaparin, 40 mg QD + Placebo: Participants received enoxaparin, 40 mg QD subcutaneously, and matching apixaban-placebo tablets BID
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Serious Adverse Events (participants affected / at risk) | 184/2673 | 172/2659
Other Adverse Events (participants affected / at risk) | 1260/2673 | 1315/2659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban, 2.5 mg BID + Placebo (N=2673) | Enoxaparin, 40 mg QD + Placebo (N=2659)
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 4 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Localised infection (Infections and infestations) | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Peroneal nerve palsy (Nervous system disorders) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Impaired healing (General disorders) | 1 | 2
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2
Tachycardia (Cardiac disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 8 | 18
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 5 | 11
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 4 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 4
Paralysis (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pyrexia (General disorders) | 3 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Wound infection (Infections and infestations) | 7 | 3
Wound secretion (Injury, poisoning and procedural complications) | 5 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Appendicitis (Infections and infestations) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Blood culture positive (Investigations) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Contrast media allergy (Immune system disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 6 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Inflammation of wound (General disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Monoparesis (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Suicide attempt (Psychiatric disorders) | 1 | 0
Unequal limb length (Musculoskeletal and connective tissue disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Vascular disorders) | 2 | 0
Aphasia (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 3
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
Body temperature increased (Investigations) | 2 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Catheter site discharge (General disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Drug level increased (Investigations) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 4
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 5 | 5
Oxygen saturation decreased (Investigations) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Postoperative wound infection (Infections and infestations) | 3 | 5
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 2 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 4 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Secretion discharge (General disorders) | 2 | 3
Sedation (Nervous system disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 3 | 7
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Ischaemia (Vascular disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 5 | 1
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bloody discharge (General disorders) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 8 | 7
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 3
Post procedural infection (Infections and infestations) | 2 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 2 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban, 2.5 mg BID + Placebo (N=2673) | Enoxaparin, 40 mg QD + Placebo (N=2659)
Procedural pain (Injury, poisoning and procedural complications) | 421 | 426
Dizziness (Nervous system disorders) | 185 | 154
Insomnia (Psychiatric disorders) | 138 | 132
Tachycardia (Cardiac disorders) | 123 | 137
Oedema peripheral (General disorders) | 156 | 141
Pyrexia (General disorders) | 236 | 242
Constipation (Gastrointestinal disorders) | 318 | 364
Hypotension (Vascular disorders) | 259 | 262
Nausea (Gastrointestinal disorders) | 485 | 529
Urinary retention (Renal and urinary disorders) | 174 | 152
Anaemia postoperative (Injury, poisoning and procedural complications) | 163 | 156
Vomiting (Gastrointestinal disorders) | 211 | 262

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.